CLINICAL TRIAL: NCT06288282
Title: Behavioral and Cognitive Predictors of Persistent Pain and Opioid Misuse in Chronic Pain
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Chinwe Nwaneshiudu, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-23-01287
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Chronic Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic back pain with lumbar, cervical or thoracic spine diagnoses.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention will be used.

SUMMARY:
Chronic lower back pain (CLBP) affects approximately 20% of the global population. The study objective is to determine if impulsivity, inhibitory control, drug choice, and/or cognitive distortions predict opioid misuse and disability in patients with chronic pain. This is a prospective consented cross-sectional study characterizing behavioral and cognitive phenotypes using both patient-reported survey measures and cognitive testing. Outcome measures include correlations between impulsivity measures, opioid drug choice responses and cognitive distortion scores, and risk for opioid misuse (Primary outcomes: COMM scores, SOAPPR scores). Secondary outcomes is BPI measurement. A Certificate of Confidentiality will provide additional protections for participants.

ELIGIBILITY:
Inclusion Criteria:

* With diagnoses related to chronic lower back pain
* Age above 18yrs
* Non pregnant

Exclusion Criteria:

* Cancer pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: chronic back pain
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Screener and Opioid Assessment for patients with pain revised (SOAPPR) | within 12 months
  Risk of opioid misuse with the Screener and Opioid Assessment for Patients with Pain Revised (SOAPPR). The Screener and Opioid Assessment for Patients with Pain-Revised (SOAPP-R) is a 24-item self-report questionnaire with total scores ranging from 0 to 24 that is used to predict risk of aberrant medication-related behaviors among chronic pain patients, with higher scores indicating higher risk of aberrant behaviors.
Current Opioid misuse measure (COMM) surveys | within 12 months
  Current opioid misuse measures with the Current Opioid misuse measure (COMM) surveys. The COMM is a 17-item self-report measure with total scores ranging from 0 to 68 that is used to identify risk of opioid misuse among chronic pain patients, with higher scores indicating higher risk of opioid misuse.

SECONDARY OUTCOMES:
Pain Intensity with Brief Pain inventory (BPI) | within 12 months
  The Brief Pain Inventory (BPI) pain intensity scale is a 0 to 10 numeric rating scale used to assess a patient's pain intensity, with 0 being no pain and 10 being pain as bad as you can imagine. Higher scores indicate higher pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Chinwe Nwaneshiudu, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Pain management centers, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: SAP, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis.
  Proposals should be directed to chinwe.nwaneshiudu@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third-party website (TBD)